CLINICAL TRIAL: NCT02566330
Title: The Effect of the EndoBarrier Device: A 3-year Follow up of a Randomized Clinical Trial
Brief Title: The EndoBarrier Device: A 3-year Follow up Study
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Selwyn van Rijn, MD, Maastricht University Medical Center
Other Study IDs: NL51074.068.14
Record Dates: First submitted 2015-07-15; First posted 2015-10-02 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Obesity; Diabetes
Keywords: EndoBarrier; Duodenojejunal Bypass Liner
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- EndoBarrier: Participants who were previously enrolled in the randomized clinical EndoBarrier procedure trial at the MUMC and the Atrium Medical Centre Heerlen.
  Interventions: Device: EndoBarrier

INTERVENTIONS:
Device: EndoBarrier — The device is a 60-cm long, impermeable plastic sleeve that is open at both sides so food can pass through. The sleeve is anchored in the duodenal bulb and extends partially into the jejunum. This way the pancreatic and bile juices will only mix with the food after the sleeve, hereby creating a functional bypass of the duodenum and the proximal jejunum, which causes malabsorption of nutrients.

SUMMARY:
The aim in the current proposal is to evaluate the long-term outcome of the EndoBarrier device. The group of participants the investigators want to study participated in earlier studies at the Maastricht University Medical Center (MUMC) and the Atrium Medical Center in Heerlen. Three years of follow-up after the EndoBarrier device is now available. The investigators hope to give new insights in the postoperative status and postoperative symptoms experienced by the study participants using standardised questionnaires and evaluating blood samples. The goal of the investigators is to study the long-term effect of the EndoBarrier procedure and to possibly provide insight in the relation between success/failure and objective parameters.

DETAILED DESCRIPTION:
In this observational follow-up study of a randomised clinical trial a maximum of 29 study participants may be included. These study participants were previously enrolled in the EndoBarrier device study at the MUMC or the Atrium Medical Centre Heerlen. The focus of this study lays on the long-term outcomes measured by EWL, postoperative blood sampling and questionnaires. These measurements, samples and questionnaires will be taken to assess the long-term effectiveness of the EndoBarrier device in the treatment of morbid obesity. Participants who were previously enrolled in the EndoBarrier device study at the MUMC or at the Atrium Medical Centre in Heerlen and who have agreed to participate in this study will be requested to arrive at the outpatient clinic of the MUMC after an overnight fast. Blood sample will be taken for total cholesterol, HDL, LDL, triglycerides, Hb, Ht, iron, HbA1c, insulin levels, glucose, amylase, lipase, C-peptide, Creatinine, vitamin D, Calcium, ALAT, ASAT, AF, gamma GT, albumin, CK-18, L-FABP, FGF19, Total bile salts and bile salt composition. These parameters are associated with risk factors in morbid obesity namely: Nonalcoholic Fatty Liver disease, hypertension, diabetes mellitus type II (DMII), coronary heart disease and osteoarthritis. After the blood sampling, physical health will be assessed by means of standard physical examination (weight, waist size, length, blood pressure, heart rate, breathing frequency). Then, the participant will be requested to fill in a validated questionnaire. In this study the SF-36 quality of life questionnaire will be used. This is a validated questionnaire assessing non-specific symptoms and quality of life after Bariatric surgery.

Three years of follow-up after the EndoBarrier device is now available. The investigators hope to give new insights in the postoperative status and postoperative symptoms experienced by participants using standardised questionnaires and evaluating blood samples. The goal of the investigators is to study the long-term effect of the EndoBarrier procedure and to possibly provide insight in the relation between success/failure and objective parameters.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were previously enrolled in the randomized clinical EndoBarrier procedure trial at the MUMC and the Atrium Medical Centre Heerlen regardless of their excess weight loss.
* Participants who have a follow up of at least 3 years.
* Signed informed consent.

Exclusion Criteria:

* Post-EndoBarrier conventional bariatric surgery
* Participants who were lost to follow-up during the previous conducted EndoBarrier clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this observational follow-up study of a randomized clinical trial a maximum of 29 participants may be included who were previously enrolled in the EndoBarrier device study at the MUMC or the Atrium Medical Centre Heerlen.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Excess Weight (%) | 36 months post explant EndoBarrier Liner

SECONDARY OUTCOMES:
Insulin levels (mmol/L) | 36 months post explant EndoBarrier Liner
Total Cholesterol (mmol/L) | 36 months post explant EndoBarrier Liner
SF-36 health related quality of life, patient-reported survey of patient health | 36 months post explant EndoBarrier Liner
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
FGF 19 (ng/ml) | 36 months post explant EndoBarrier Liner
ASAT (U/L) | 36 months post explant EndoBarrier Liner
Amylase (U/L) | 36 months post explant EndoBarrier Liner
Systolic blood pressure (mmHg) | 36 months post explant EndoBarrier Liner
BMI (Kg/M2) | 36 months post explant EndoBarrier Liner
Diastolic blood pressure (mmHg) | 36 months post explant EndoBarrier Liner
glucose levels (mmol/L) | 36 months post explant EndoBarrier Liner
HbA1c level (%) | 36 months post explant EndoBarrier Liner
Triglycerides (mmol/L) | 36 months post explant EndoBarrier Liner
HDL (mmol/L) | 36 months post explant EndoBarrier Liner
LDL (mmol/L) | 36 months post explant EndoBarrier Liner
L-FABP (ng/ml) | 36 months post explant EndoBarrier Liner
Lipase (U/L) | 36 months post explant EndoBarrier Liner
ALAT (U/L) | 36 months post explant EndoBarrier Liner
AF (U/L) | 36 months post explant EndoBarrier Liner
GammaGT (U/L) | 36 months post explant EndoBarrier Liner
Albumin (g/L) | 36 months post explant EndoBarrier Liner
CK-18 (U/L) | 36 months post explant EndoBarrier Liner
C-peptide (nmol/L) | 36 months post explant EndoBarrier Liner

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Bouvy, MD, PhD, Principal Investigator — Maastricht University Medical Center, The Netherlands
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands